CLINICAL TRIAL: NCT06177665
Title: Comparison of Erector Spina Plan Block and Rhomboid Intercostal Block for Postoperative Pain Managment in Patients Undergoing Unilateral Breast Surgery
Brief Title: Comparison of Erector Spina Plan Block and Rhomboid Intercostal Block in Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Gulnihal Avci, Doctor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: KAEK/08.bI.02
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Pain; Analgesia
Keywords: Regional Anesthesia; Erector Spinae Plane Block; Rhomboid Intercostal Block; Breast Surgery
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erector Spinae Plane Block (Experimental): Ultrasound(US)-guided erector spinae plan block(ESP) with 20 ml 0,25% bupivacaine at T4 vertebra level will performe preoperatively to all patients in the ESP group.
  Interventions: Other: Erector Spinae Plane Block
- Rhomboid Intercostal Block (Experimental): Ultrasound(US)-guided rhomboid intercostal block(RIB) with 20 ml 0,25% bupivacaine at T5-T6 vertebra level will performe preoperatively to all patients in the RIB group.
  Interventions: Other: Rhomboid Intercostal Block

INTERVENTIONS:
Other: Erector Spinae Plane Block — Ultrasound(US)-guided erector spinae plan block(ESP) with 20 ml 0,25% bupivacaine at T4 vertebra level will performe preoperatively to all patients in the ESP group.
  Arms: Erector Spinae Plane Block
Other: Rhomboid Intercostal Block — Ultrasound(US)-guided rhomboid intercostal block(RIB) with 20 ml 0,25% bupivacaine at T5-T6 vertebra level will performe preoperatively to all patients in the RIB group.
  Arms: Rhomboid Intercostal Block

SUMMARY:
In this study, the investigators compared ultrasound-guided erector spinae plane (ESP) block and rhomboid intercostal block (RIB) on postoperative analgesic effect in unilateral breast surgery.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, written consent was obtained from all patients.Patients who meet eligibility requirements will be randomized in a 1:1 ratio to erector spinae plane block and rhomboid intercostal block.

ELIGIBILITY:
Inclusion Criteria

* Patients who will undergo unilateral breast-conserving surgery (BCS) or modified radical mastectomy (MRM) with or without axillary lymph node dissection
* Patients undergoing elective surgery
* ASA (American Society of Anesthesiologists) physical status classification I-III

Exclusion Criteria:

* Use of anticoagulants
* Allergy to the medications to be used
* Patients who use analgesic drugs due to a history of chronic pain
* ASA (American Society of Anesthesiologists) physical status classification IV-V
* Patients with psychiatric disorders
* Presence of infection in the area where the block will be applied
* Presence of deformity in the patient's spinal, paraspinal and area where the block will be applied
* The patient does not accept the block application or cannot cooperate with the patient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Morphin Consumption | during postoperative 24 hours
  Patients in both groups will provide with intravenous patient-controlled analgesia device containing morphine for postoperative analgesia

SECONDARY OUTCOMES:
Numerical Rating Scale(NRS) | during postoperative 24 hours
  A numerical rating scale(NRS) requires the patient to rate their pain on defined scale.For example , 0-10 where 0 is no pain and 10 is the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Sevim Cesur Okan, Study Director — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

REFERENCES:
- See also: Comparison of rhomboid intercostal nerve block, erector spinae plane block and serratus plane block on analgesia for modified radical mastectomy: A prospective randomised controlled trial. — https://pubmed.ncbi.nlm.nih.gov/34133831/
- See also: Rhomboid intercostal block — https://pubmed.ncbi.nlm.nih.gov/27291611/
- See also: Ultrasound-guided fascial plane blocks of the chest wall: a state-of-the-art review — https://pubmed.ncbi.nlm.nih.gov/33426660/